CLINICAL TRIAL: NCT01830127
Title: A Phase IIb Open Label Study of BI 207127 in Combination With Faldaprevir and Ribavirin in Patients With Moderate Hepatic Impairment (Child-Pugh B) With Genotype 1b Chronic Hepatitis C Infection
Brief Title: BI 207127 / Faldaprevir Combination Therapy in Hepatic Impairment (Child-Pugh B) Patients With Genotype 1b Chronic Hepatitis C Infection: HCVerso3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1241.30; 2012-003534-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-03-22; First posted 2013-04-12 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; deleobuvir; faldaprevir

ARMS (2):
- cohort A CPA (Experimental): Cohort A CPA BI 207127/QD Faldaprevir Ribavirin
  Interventions: Drug: Ribavirin; Drug: Faldaprevir; Drug: BI 207127 low dose
- cohort A CPB (Experimental): Cohort B CPB BI 207127/QD Faldaprevir Ribavirin
  Interventions: Drug: BI 207127 high dose; Drug: Ribavirin; Drug: Faldaprevir

INTERVENTIONS:
Drug: Ribavirin — 24 Weeks
  Arms: cohort A CPA
Drug: BI 207127 high dose — 24 Weeks
  Arms: cohort A CPB
Drug: Faldaprevir — 24 Weeks
  Arms: cohort A CPA
Drug: Ribavirin — 24 Weeks
  Arms: cohort A CPB
Drug: BI 207127 low dose — 24 Weeks
  Arms: cohort A CPA
Drug: Faldaprevir — 24 Weeks
  Arms: cohort A CPB

SUMMARY:
To assess the pharmacokenetic characteristics of 600 mg BID BI 207127 / 120 mg QD faldaprevir /ribavirin in a small number of GT1b HCV infected patients with mild hepatic impairment (CPA) (Arm 1) versus 400 mg BID BI 207127 / 120 mg QD faldaprevir /ribavirin in a small number of GT1b HCV infected patients with moderate hepatic impairment (CPB) (Arm 2).

ELIGIBILITY:
Inclusion criteria:

1. Treatment naïve and treatment experienced patients (prior relapse, interferon intolerant, and [allowed in Cohort A only] prior partial response).
2. Chronic HCV infection of genotype 1 (GT1), sub-GT1b virus only.
3. Liver cirrhosis defined as Metavir Grade=4 or Ishak Grade =5 on liver biopsy or liver stiffness of =13 kPa on fibroscan.

Exclusion criteria:

1. HCV infection of mixed genotype (1/2, 1/3, and 1/4) or mixed sub-GT1a/1b or undefined diagnosed by genotypic testing at screening
2. Liver disease due to causes other than chronic HCV infection which may include but is not limited to hemochromatosis, Wilson's disease, or autoimmune liver diseases.
3. HIV infection
4. Patients who have been previously treated with an investigational or approved DAA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- United States (6):
  - 1241.30.10003 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1241.30.10007 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1241.30.10001 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1241.30.10012 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 1241.30.10011 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1241.30.10002 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
- Germany (8):
  - 1241.30.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.30.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.30.49005 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.30.49008 Boehringer Ingelheim Investigational Site, Bonn
  - 1241.30.49006 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1241.30.49001 Boehringer Ingelheim Investigational Site, Hanover
  - 1241.30.49003 Boehringer Ingelheim Investigational Site, Leipzig
  - 1241.30.49007 Boehringer Ingelheim Investigational Site, Mainz
- Spain (4):
  - 1241.30.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.30.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.30.34003 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.30.34001 Boehringer Ingelheim Investigational Site, Majadahonda (Madrid)
- 1241.30.44002 Boehringer Ingelheim Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Sarrazin C, Manns M, Calleja JL, Garcia-Samaniego J, Forns X, Kaste R, Bai X, Wu J, Stern JO. HCVerso3: An Open-Label, Phase IIb Study of Faldaprevir and Deleobuvir with Ribavirin in Hepatitis C Virus Genotype-1b-Infected Patients with Cirrhosis and Moderate Hepatic Impairment. PLoS One. 2016 Dec 28;11(12):e0168544. doi: 10.1371/journal.pone.0168544. eCollection 2016. PMID 28030579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 patients were enrolled and treated with Deleobuvir (DBV) / Faldaprevir (FDV) / Ribavirin (RBV): 18 patients with Child-Pugh A (mild hepatic impairment) and 17 patients with Child-Pugh B (moderate hepatic impairment).
Pre-assignment Details: This was phase IIb open label study of BI 207127 (Deleobuvir) in combination with faldaprevir and ribavirin in patients with mild hepatic impairment (Child-Pugh A) and moderate hepatic impairment (Child-Pugh B) with genotype 1b chronic hepatitis C infection.
Groups:
- Arm1: Child-Pugh A: Arm 1 (genotype 1b) - 600mg DBV tablet taken orally twice daily (BID) plus 120mg FDV capsule taken orally once daily (QD) plus RBV tablet taken orally twice daily for 24 weeks.
- Arm2: Child-Pugh B: Arm 2 (genotype 1b) - 400mg DBV tablet taken orally twice daily (BID) plus 120mg FDV capsule taken orally once daily (QD) plus RBV tablet taken orally twice daily for 24 weeks.
Period: Overall Study
Arm/Group | Arm1: Child-Pugh A | Arm2: Child-Pugh B
Started | 18 | 17
Completed | 13 | 8
Not Completed | 5 | 9
Not completed — Adverse Event | 1 | 6
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other reason not defined above | 0 | 2

BASELINE CHARACTERISTICS:
Population: (Treated Set) All patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment, regardless of randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm1: Child-Pugh A | Arm2: Child-Pugh B | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (8.8) | 56.6 (9.7) | 57.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: SVR12: Plasma HCV RNA Level Less Than 25 IU/mL at 12 Weeks After End of Treatment (EOT)
Description: Sustained virologic response (SVR) at Week 12 post-treatment (SVR12): Plasma Hepatitis C virus Ribonucleic acid (HCV RNA) level <25 IU/mL(international units per millilitre) at 12 weeks after EOT. SVR12 was analyzed in a descriptive manner using percentage.
Time Frame: 12 weeks after End of Treatment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm1: Child-Pugh A | Arm2: Child-Pugh B
Number analyzed (Participants) | 18 | 17
Percentage of participants | 61.1 [38.6 to 83.6] | 52.9 [29.2 to 76.7]

2. Secondary Outcome: SVR4: Plasma HCV RNA Level Less Than 25 IU/mL at 4 Weeks After End of Treatment (EOT)
Description: Sustained virologic response (SVR) at Week 4 post-treatment (SVR4): Plasma Hepatitis C virus Ribonucleic acid (HCV RNA) level <25 IU/mL at 4 weeks after EOT. SVR4 was analyzed in a descriptive manner using percentage.
Time Frame: 4 weeks after End of Treatment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm1: Child-Pugh A | Arm2: Child-Pugh B
Number analyzed (Participants) | 18 | 17
Percentage of participants | 72.2 [51.5 to 92.9] | 76.5 [56.3 to 96.6]

ADVERSE EVENTS:
Time Frame: From first drug administration until last drug administration plus 28 days, up to 28 weeks.
Arm/Group | Arm1: Child-Pugh A | Arm2: Child-Pugh B
Serious Adverse Events (participants affected / at risk) | 1/18 | 9/17
Other Adverse Events (participants affected / at risk) | 17/18 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1: Child-Pugh A (N=18) | Arm2: Child-Pugh B (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 3
Peritonitis bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm1: Child-Pugh A (N=18) | Arm2: Child-Pugh B (N=17)
Anaemia (Blood and lymphatic system disorders) | 6 | 8
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Erythema of eyelid (Eye disorders) | 1 | 0
Ocular icterus (Eye disorders) | 6 | 3
Photophobia (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 7
Cheilitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 9 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Faeces soft (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 13
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 6
Asthenia (General disorders) | 7 | 7
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 3
Gait disturbance (General disorders) | 1 | 2
Mucosal dryness (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 4 | 5
Pyrexia (General disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 4
Jaundice (Hepatobiliary disorders) | 5 | 8
Bronchitis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hepatitis C RNA increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Waist circumference increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 5
Dysgeusia (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypertonia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 1
Parosmia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 4
Libido increased (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Vasospasm (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Because the company decided to stop the DBV development program, analyses for this trial were limited to the basic requirement for efficacy, and only the primary endpoint and secondary endpoint were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.